CLINICAL TRIAL: NCT05674838
Title: Evaluation of the Use of Leg Elevation on a Peanut Ball to Prevent Hypotension Following Epidural Anesthesia in Laboring Women
Brief Title: Leg Elevation to Prevent Hypotension During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-045
Record Dates: First submitted 2022-12-21; First posted 2023-01-09 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hypotension; Labor Complication
MeSH Terms: conditions — Hypotension; Obstetric Labor Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention - Leg Elevation Arm (Experimental): Immediately after epidural placement, patient will be placed in a left tilt position with her hip on a wedge and both of her legs elevated on an orange peanut ball. She will remain in this position for approximately 40 minutes.
  Interventions: Other: Leg Elevation
- Control - No Leg Elevation Arm (No Intervention): Immediately after epidural placement, patient will be placed in a left tilt position with her hip on a wedge. She will remain in this position for approximately 40 minutes.

INTERVENTIONS:
Other: Leg Elevation — Immediately after epidural placement, patient will be placed in a left tilt position with her hip on a wedge and both of her legs elevated on an orange peanut ball. She will remain in this position for approximately 40 minutes.
  Arms: Experimental Intervention - Leg Elevation Arm

SUMMARY:
When hypotension is related to epidural placement, this can occur within 15-60 minutes after placement. The purpose of this study is to build upon this preliminary work and to use a randomized controlled trial to examine the effectiveness of leg elevation in preventing hypotension among a larger sample of laboring women who receive an epidural analgesia. This study will use a randomized, non-blinded, controlled design with two arms:

Arm 1: Patient will be put in a left tilt position with her hip on a wedge and both legs elevated on a peanut ball. She'll remain in this position for approximately 40 minutes.

Arm 2: Patient will be put in a left tilt position with her hip on a wedge and no leg elevation. She'll remain in this position for approximately 40 minutes.

DETAILED DESCRIPTION:
When hypotension is related to epidural placement, this can occur within 15-60 minutes after placement. The purpose of this study is to build upon this preliminary work and to use a randomized controlled trial to examine the effectiveness of leg elevation in preventing hypotension among a larger sample of laboring women who receive an epidural analgesia. This study will use a randomized, non-blinded, controlled design with two arms:

Arm 1: Patient will be put in a left tilt position with her hip on a wedge and both legs elevated on a peanut ball. She'll remain in this position for approximately 40 minutes.

Arm 2: Patient will be put in a left tilt position with her hip on a wedge and no leg elevation. She'll remain in this position for approximately 40 minutes.

Outcome variables include occurrence of maternal hypotension or late or prolonged decelerations within the first hour after epidural placement.

ELIGIBILITY:
Inclusion Criteria:

* Laboring at Good Samaritan Hospital Labor & Delivery Unit
* 37+ weeks gestation
* Planned vaginal delivery
* Planned epidural analgesia

Exclusion Criteria:

* Under 18 years old
* Does not speak English
* Unable to consent to involvement in the research study
* Attended less than 3 prenatal care office visits
* Diagnosed with fetal demise
* Diagnosed with fetal anomalies
* Contraindications to both legs being elevated (ex: fractured bones, lower limb amputation, etc.)
* Contraindications to receiving 1L of IV fluids
* Requiring IV hypertensive medications
* Requiring IV magnesium

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Laboring women only
Enrollment: 102 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Intervention - Leg Elevation Arm | Control - No Leg Elevation Arm
Started | 58 | 44
Completed | 54 | 38
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Intervention - Leg Elevation Arm | Control - No Leg Elevation Arm | Total
Number analyzed (Participants) | 54 | 38 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years as continuous variable
  years | 30.4 (4.4) | 29.9 (4.2) | 30.2 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex as self-reported
  Participants
    Female | 54 | 38 | 92
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Maternal Hypotension Requiring Treatment
Description: SBP requiring treatment by the anesthesia provider
Time Frame: 40 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Intervention - Leg Elevation Arm | Control - No Leg Elevation Arm
Number analyzed (Participants) | 54 | 38
Participants
  Maternal Hypotension requiring Intervention | 6 | 11
  No Maternal Hypotension requiring Intervention | 48 | 27

2. Primary Outcome: Number of Patients With Late or Prolonged Decelerations on the Fetal Heart Tracings
Description: Any late or prolonged decelerations on the fetal heart tracings
Time Frame: 40 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Intervention - Leg Elevation Arm | Control - No Leg Elevation Arm
Number analyzed (Participants) | 54 | 38
Participants
  Late or Prolonged Decelerations | 10 | 12
  No Late or Prolonged Decelerations | 44 | 26

ADVERSE EVENTS:
Time Frame: from enrollment until end of delivery, up to 2 days
Arm/Group | Experimental Intervention - Leg Elevation Arm | Control - No Leg Elevation Arm
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/38
Other Adverse Events (participants affected / at risk) | 0/54 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT05674838/Prot_SAP_000.pdf